CLINICAL TRIAL: NCT04059939
Title: Evidence-Based Interventions to Enhance Outcomes Among Struggling Readers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Amie E. Grills, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHD087706A
Record Dates: First submitted 2017-02-09; First posted 2019-08-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Reading Disability; Anxiety
MeSH Terms: conditions — Dyslexia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants and evaluators are not told which interventions individual participants have been assigned to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reading Plus Attention Control (Experimental)
  Interventions: Other: Reading; Other: Attention Control (math practice)
- Reading Plus Anxiety (Experimental)
  Interventions: Other: Reading; Behavioral: Anxiety Management
- BAU (Active Comparator)
  Interventions: Other: Classroom Business as Usual

INTERVENTIONS:
Other: Reading — Small group reading instruction
  Arms: Reading Plus Anxiety; Reading Plus Attention Control
Behavioral: Anxiety Management — small group anxiety management skills instruction
  Arms: Reading Plus Anxiety
Other: Classroom Business as Usual — Classroom Business as Usual
  Arms: BAU
Other: Attention Control (math practice) — Attention Control (math practice)
  Arms: Reading Plus Attention Control

SUMMARY:
Despite decades of research on reading disabilities, little is known about improving reading in the middle grades (i.e., grades 3-6) and advancements have been hindered by the narrow focus on reading problems alone without acknowledgement of non-academic factors shown to affect learning (e.g., child self-regulation). This proposal employs a highly innovative approach aimed at improving intervention outcomes through the integration of evidence-based practices for addressing reading, as well as self-regulation/socioemotional skills, difficulties known to occur in a substantial percentage of struggling readers and to negatively influence academic performance. This project represents translational research that directly informs the practice community (schools, clinicians, teachers, parents), by identifying novel instructional practices that can be aggregated to more effectively influence student outcomes and reduce disparities in academic and socioemotional domains.

DETAILED DESCRIPTION:
While considerable knowledge has been accumulated on improving reading for students with reading disabilities in the primary grades, reading interventions conducted with middle-grades (i.e., grades 3-6) have been rare and have typically evidenced low impacts, even when more intensive interventions are provided for increasingly longer durations. One hindrance to extant interventions has been the narrow focus on reading problems without addressing non-academic (e.g., self-regulation, socioemotional) factors known to also affect learning. Thus, investigations of the efficacy derived from integrating additional components into standard reading skills interventions are necessary. Anxiety represents a particularly salient target for such an approach, as it is among the most commonly reported mental health issues of childhood, and significant associations have been found between anxiety and academic outcomes. Further, an overwhelming number of children who are struggling to read or who fail to respond to reading interventions report elevated anxiety. The purpose of this proposal is to evaluate an integrated program designed for middle-grade readers and comprised of evidence-based practices for the treatment of anxiety and reading difficulties. A pilot study of this program, conducted with 36 students randomized to treatment and control conditions, demonstrated its feasibility and positive effects on anxiety outcomes. The RCT will extend this work by comparing the combined reading and anxiety intervention with a reading-only condition and a control condition. Struggling readers will be included in this study and will receive two years of intervention. The study will assess efficacy of the interventions at reducing anxiety and improving reading at post-intervention and 6-month follow-up (Aim 1). This project significantly enhances extant research on interventions for struggling reading by examining mechanisms of action associated with augmented outcomes among students who receive the combined intervention (Aim 2), and by determining potential moderators of intervention effects (Aim 3). In all, between 300 and 350 ethnically diverse students will be recruited. A multi-informant (student, parent, teacher), multi-method (e.g., survey, standardized test, experiential sampling) assessment will be used. Relevance of this project lies in the determination of whether the inclusion of anxiety management skills enhances existing intervention outcomes for struggling readers in the upper elementary grades (concurrently/longitudinally). Examination of contextual and mitigating factors are further relevant for understanding the complex etiology of response to intervention among struggling readers. This project represents translational research that directly informs the practice community (e.g., clinicians, teachers) by identifying novel instructional practices that can be aggregated to more effectively influence student outcomes. By providing socioemotional skills training with a reading intervention using a school-based delivery model, this work has the potential of reducing disparities in mental health outcomes by reaching students of diverse backgrounds (e.g., ethnicity, SES) who would be otherwise less likely to receive such services.

NOTE: The Covid-19 pandemic emerged mid-project and altered several of our plans for this project, as well as led to a mid-project extension. Specifically, this was designed as a 2-cohort, multi-year intervention study. While Cohort 1 completed all planned milestones and activities, for Cohort 2 the intervention was ongoing when the pandemic closed all schools. A third Cohort was then added when schools reopened, but students in Cohort 3 only received 1 year of the intended 2-year intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 3rd or 4th grade
* Demonstrate difficulty with reading (which is defined as scoring at or below a standard score of 90 on the Gates MacGinite Reading Comprehension Test
* Difficulty with reading must be confirmed by classroom teacher/school

Exclusion Criteria:

* Students with limited English proficient (due to all assessments being administered in English only)
* Students in life skills classes (due to task appropriateness)
* Students who have an unrelated neurological disorder (e.g., tumor, traumatic brain injury)
* Students who have a severe psychiatric disorder that prevents assessment (e.g., autism), or who have an uncorrected sensory disorder

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 542 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Test of Word Reading Efficiency | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Measures "ability to pronounce printed words and phonemically regular nonwords accurately and fluently"
Multidimensional Anxiety Scale for Children | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
  39-item scale of anxiety comprised of four subscales: Physical Symptoms, Harm Avoidance, Social Anxiety, and Separation/Panic. Response options range from 0-3. A total score is comprised of all subscales added together. The total score can range from 0-117. The range of the subscales are as follows: Physical Symptoms (0-36), Harm Avoidance (0-27), Social Anxiety (0-27), Separation/Panic (0-27). Higher scores indicate more anxiety. There are child, parent, teacher versions of this scale.
Woodcock-Johnson Psycho-Educational Test Battery-III | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Two subtests: Letter-Word Identification and Word Attack. Scores are reported as standard scores in a range of 0-200+ or percentile ranks in a range of 0.1 to 99.9. The higher the score the greater the achievement level of the student.

SECONDARY OUTCOMES:
Children's Test Anxiety Scale | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
  30-item scale with a 4-point Likert Scale (1-4). Scale ranges from 30-120 with higher scores indicating greater test anxiety.
Reading Anxiety Scale | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
  6-item scale adapted from the Wigfield and Meece (1988) Math Anxiety Scale. Designed to assess worries and stressed feelings about reading instruction and reading tests. Participants responded to each item with a 5-point Likert Scale from Never to Always. Higher scores indicate greater levels of reading anxiety.
Attention | Change from baseline to post-intervention year 1, Change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  child attention scale, Effortful Control-Persistence/Low Distractibility subscale, Strength and Weaknesses of Attention-Deficit/Hyperactivity Disorder, (SWAN) parent/teacher reported attention
Test of Silent Word Reading Efficiency and Comprehension | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
Dynamic Indicators of Basic Early Literacy Skills | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Oral Reading Fluency
Beck Anxiety Inventory | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
  Self-report measure of anxiety in the past month. 21-item scale with a 4-point Likert scale. from 0-3. Items summed together. Scale range from 0-63. Score of 0-21= low anxiety. Score of 22-35 = moderate anxiety. Score of 36 and above = potentially concerning levels of anxiety. Administered to parents. Administered to intervention teachers in cohorot 2.
Beck Youth Inventories (BYI) | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, BYI depression subscale was not administered at post-intervention Y1
  Self-report measure comprised of five inventories, which measure depression, anxiety, anger, disruptive behavior, and self-concept. Each inventory has 20-items which are scored on a 4-point Likert scale (0-3). Higher scores indicate greater amounts of concept (i.e., depression, anxiety, anger, disruptive behavior, and self-concept) being measured.
Stress management skills evaluation | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
Confusion, Hubbub, and Order Scale (CHAOS Survey) | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3
  15-items with a 4-point Likert Scale (1-4) measuring the home environment. Completed by parent/caregiver. Total score is created by summing the responses to the items. Range is 15-60. Higher scores indicate more chaotic home environments.
Reading Comprehension | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Kaufman Test of Educational Achievement-III (KTEA-3)
Fluency/Comprehension | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Test of Silent Word Reading Fluency
Verbal Knowledge/Matrices | Change from baseline to post-intervention year 1, change from baseline to post-intervention year 2, change from year 1 to year 2, change from year 2 to year 3; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Kaufman Brief Intelligence Test
Math Calculation | Change from baseline to post-intervention year 2
  Woodcock-Johnson Psycho-Educational Test Battery-III Calculation
Essential Word Knowledge | Change from baseline to post-intervention year 2
Reading Comprehension | Change from post-intervention year 1 to post-intervention year 2; In cohort 2, same time frames, except it was not administered at post-intervention Y1
  Gates-MacGinitie Reading Comprehension
Home Literacy Questions | Cohort 2 Only- administered at post-intervention Y1
  A total of 7 questions (e.g., how many children's books are in your home; how many times per a week have you read with your child while schools have been closed?) examine home literacy prior to COVID19 and during COVID19.

CONTACTS AND LOCATIONS:
Overall Officials: Amie E Grills, PhD, Principal Investigator — Boston University; Sharon Vaughn, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No